CLINICAL TRIAL: NCT06279455
Title: Evaluation of the Effect of Pelvic Floor Muscle Exercise During Pregnancy on Sexual Function, Lower Urinary Tract Symptoms and Birth Process
Brief Title: Pelvic Floor Muscle Exercise During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Zahide Celebi, M.Sc./Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-74555795-050.01.04-392120
Record Dates: First submitted 2023-12-28; First posted 2024-02-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Lower Urinary Tract Symptoms; Sexual Function
Keywords: Lower Urinary Tract Symptoms; Pelvic Floor Muscle Exercise; Pregnancy; Sexual Function; Birth Process
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Pelvic Floor Muscle Exercise Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Pregnant women in the control group were not trained and routine follow-up was performed in the outpatient clinic.
  Female Sexual Function Index (FSFI) and International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms Long Form (ICIQ-FLUTS LF) at 18-20 weeks of gestation, Mid-term Evaluation Form at 26 weeks of gestation and FSFI and ICIQ-FLUTS LF at 32 weeks of gestation were applied to pregnant women in the control group participating in the study. Data on the birth process were collected between 3-7th days after birth with the Birth Process Follow-up Form.
- Experimental Group (Experimental): Two sessions of training were given using the "Pelvic Floor Health & Sexual Life in Pregnancy Training Booklet" and the pelvic floor muscle exercise training video developed by the researcher between 18-20 weeks of pregnancy. Before the training, the FSFI and the ICIQ-FLUTS LF were administered to the pregnant women. Pregnant women were asked to perform pelvic floor muscle exercises, 3 sets a day, 3 days a week, for 12 weeks, starting from the 20th week of pregnancy, and record them in the Pelvic Floor Muscle Exercise Follow-up Form created by the researcher. By scanning the literature, 1 set of exercise was determined as 8-12 slow contractions (6-8 seconds) followed by 3-4 fast contractions (1 second).
  Interventions: Other: Pelvic Floor Muscle Exercise

INTERVENTIONS:
Other: Pelvic Floor Muscle Exercise — A 12-week pelvic floor muscle exercise program was applied to pregnant women.
  Arms: Experimental Group

SUMMARY:
This study was conducted to evaluate the effects of pelvic floor muscle exercises during pregnancy on sexual function, lower urinary tract symptoms and birth process. The research was conducted with pregnant women who applied to the Pregnancy Outpatient Clinic of Istanbul University-Cerrahpasa Cerrahpasa Faculty of Medicine Hospital. Power analysis was performed to determine the number of samples to be included in the study. It was determined that 29 pregnant women should be included in each group (experimental and control). Considering the possibility of data loss, 50 pregnant women were included in each group. As a result of the exclusion of 8 women who withdrew from participating in the study, 5 women due to risky pregnancies (bleeding, preeclampsia and gestational diabetes) and 17 women due to cesarean delivery, the data of 35 pregnant women in the experimental group and 35 pregnant women in the control group were obtained. Pregnant women in the experimental group were gestational aged 18-20. Two sessions of training were given on female reproductive and urinary system anatomy, physiological changes during pregnancy and their effects on sexual life, and pelvic floor muscle exercises, using the "Pelvic Floor Health & Sexual Life Training Booklet during Pregnancy" and the pelvic floor muscle exercise training video developed by the researcher between the weeks of pregnancy. Pregnant women were asked to perform pelvic floor muscle exercises, 3 sets a day, 3 days a week, for 12 weeks, starting from the 20th week of pregnancy, and record them in the Pelvic Floor Muscle Exercise Follow-up Form created by the researcher. Pregnant women in the control group were not given any training and were routinely monitored in the outpatient clinic. Pregnant women who apply to the outpatient clinic are examined by nurses, with their vital signs taken and anamnesis taken by the physician. Recommendations are made regarding the complaints of pregnant women. Non-stress tests are routinely applied to pregnant women who are at the 36th week of pregnancy and above.

DETAILED DESCRIPTION:
Purpose of the research This study was conducted to evaluate the effects of pelvic floor muscle exercises during pregnancy on sexual function, lower urinary tract symptoms and birth process.

Type of Research This research is of randomized controlled prospective type.

Place and Time the Research The research was conducted at the Pregnancy Outpatient Clinic of Istanbul University-Cerrahpasa Cerrahpasa Faculty of Medicine Hospital, Department of Gynecology and Obstetrics, between December 2022 and October 2023.

Population and Sample of the Research The population of the research consisted of pregnant women who applied to the Pregnancy Outpatient Clinic of Istanbul University-Cerrahpasa Cerrahpasa Faculty of Medicine Hospital, Department of Gynecology and Obstetrics. G*Power (3.1.9.7) Program was used to determine the sample number of pelvic floor muscle exercise (experimental group) and control groups. The Female Sexual Function Index was taken as the main parameter in the study. As a result of the power analysis performed with α=0.05 and power of 95% (effect size: 0.7), the sample was calculated as 29 pregnant women for each group. Considering that there may be losses during the study period, it was decided to include a total of 100 pregnant women between the ages of 18-40, including the experimental group (n = 50) and the control group (n = 50).

The numbers to be included in the sample were determined using the randomization program (www.randomizer.org).

As a result of the exclusion of 8 women who withdrew from participating in the study, 5 women due to risky pregnancies (bleeding, preeclampsia and gestational diabetes) and 17 women due to cesarean delivery, the data of 35 pregnant women in the experimental group and 35 pregnant women in the control group were obtained.

Research data were collected with "Personal Information Form" (between 18-20th week of pregnancy), "Female Sexual Function Index" (between 18-20th week of pregnancy and 32nd week of pregnancy), "Mid-term Evaluation Form" (26th week of pregnancy), "International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms Long Form (ICIQ-FLUTS LF)" (between 18-20th week of pregnancy and 32nd week of pregnancy), "Birth Process Follow-up Form" (between 3-7th days after birth) and "Pelvic Floor Muscle Exercise Follow-up Form" (20-32 between weeks of pregnancy).

ELIGIBILITY:
Inclusion Criteria:

* Between the 18th and 20th weeks of gestation,
* Nulliparous and single pregnancy,
* Sexually active,
* Body mass index before pregnancy <30,
* Urinary incontinence and urinary infection are not diagnosed,
* Not having a psychiatric illness,
* The spouse does not have sexual dysfunction.

Exclusion Criteria:

* Pregnant women under 18 weeks and older than 20 weeks,
* Primiparous and multiparous,
* High-risk pregnancy (multiple pregnancy, preeclampsia, gestational diabetes, pregnancy with assisted reproductive techniques),
* Pregnant women who are scheduled for elective cesarean section,
* Those who give birth by cesarean section.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Sexual Function | 12 weeks
  The outcome is sexual function of pregnant women. It will be measured with FSFI.
Lower Urinary Tract Symptoms | 12 weeks
  The outcome is lower urinary tract symptoms of pregnant women. It will be measured with ICIQ-FLUTS LF.
Birth Process | 18 weeks
  The outcome is birth outcomes. It will be evaluated with Birth Process Follow-up Form.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No